CLINICAL TRIAL: NCT02514330
Title: Concurrent Effect of Running in Different Slopes on Power Performance
Brief Title: Running Slopes and Power Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: UGF 02
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: Drop Jump; High Intensity Interval Training; Muscle Fatigue; Aerobic Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interval Training at 1% incline (Experimental): Procedure: Initial Drop Jump (20;30;40 cm), Six Stimulus of High Intensity Interval Training at 1% incline, Final Drop Jump (20;30;40 cm)
  Interventions: Other: Interval Training at 1% incline
- Interval Training at 10% incline (Experimental): Procedure: Initial Drop Jump (20;30;40 cm), Six Stimulus of High Intensity Interval Training at 10% incline, Final Drop Jump (20;30;40 cm)
  Interventions: Other: Interval Training at 10% incline
- Control (No Intervention): Procedure: Initial Drop Jump (20;30;40 cm), 20 min Rest, Final Drop Jump (20;30;40 cm)

INTERVENTIONS:
Other: Interval Training at 1% incline — Six stimuli were performed to exhaustion. The vertical drop jump strategy (height and kinematics) served to establish the magnitude of the concurrent effect
  Other Names: HIIT at 1%; High Intensity Interval Training at 1%
  Arms: Interval Training at 1% incline
Other: Interval Training at 10% incline — Six stimuli were performed to exhaustion. The vertical drop jump strategy (height and kinematics) served to establish the magnitude of the concurrent effect.
  Other Names: HIIT at 10%; High Intensity Interval Training at 10%
  Arms: Interval Training at 10% incline

SUMMARY:
The objective of the present study was to determine the effect of interval session running at high intensity with 1% or 10% gradient on the height of the drop jump. The cinematic variables concentric phase, eccentric and contact time were compared after the running session in both conditions in order to explain possible changes in the jump performance. The investigators theorize that the lower eccentric overload in the running to 10% inclination promotes higher deleterious effect on power performance of the lower limbs

DETAILED DESCRIPTION:
Physical training programs are typically composed of activities directed to the development of different valences usually stimulated in the same session. When aerobic activities of long duration prior isokinetic strength exercises, isotonic, or explosive, deleterious effects seem to be induced on performance of these valences. These short and long-term changes in muscle strength and power would be directly associated with repetitive eccentric loads that characterize the endurance running. Gradual increases in the running slope were inversely associated with a proportional reduction in the eccentric loads, which in turn would result in less muscle damage to intra and extrafusal fibers. So, the change in the slope of the race would emerge as an optional way to neutralize the competitive effect on the power performance. The research consisted of five visits. At the initial visit was conducted familiarization to vertical drop jump, and immediately after, the determination of VO2max values and their associated speed (vVO2max). The second visit was a new familiarization for the vertical drop jump followed immediately determining the Time to exhaustion performance in vVO2max (100% of VO2Max). Two jumps were performed on each of the three selected heights (20, 30 and 40 cm) were used in the experimental sessions and control only the height associated with the highest performance. In subsequent visits (third to fifth), participants performed three maximum jumps before and about 10 min after the following conditions: high intensity Interval running a 10% gradient (C10%), 1% grade (C1%) and control condition (CON).

ELIGIBILITY:
Inclusion Criteria:

* age: 18 at 45 years
* no cardiovascular or metabolic problems
* minimum level of aerobic activity recommended by American College of Sports Medicine

Exclusion Criteria:

* no joint or muscle injuries
* no use ergogenic or anabolic resources

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Kinematic of Height Jump | up to 1 month
  the same group (N=25) of subjects performed the experimental procedure in the last three sessions aiming to achieve the highest performance in all three conditions

SECONDARY OUTCOMES:
Kinematic of Concentric Phase | up to 1 month
  the same group of subjects performed the experimental procedure in the last three sessions
Kinematic of Excentric Phase | up to 1 month
  the same group of subjects performed the experimental procedure in the last three sessions
Kinematic of Contact Time | up to 1 month
  the same group of subjects performed the experimental procedure in the last three sessions

CONTACTS AND LOCATIONS:
Overall Officials: Tony Santos, Doctor, Study Director — Universidade Federal de Pernambuco